CLINICAL TRIAL: NCT04545476
Title: Novel Biomaterial Containing Gelatin, Manuka Honey, and Hydroxyapatite Enhanced Secondary Intention Healing vs. Standard Secondary Intention Healing in Mohs Surgical Defects on the Head and Distal Lower Extremities - A Randomized Clinical Trial
Brief Title: Enhanced Secondary Intention Healing vs. Standard Secondary Intention Healing in Mohs Surgical Defects on the Head and Distal Lower Extremities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Karen Arnaud, Dermatology Resident Physician, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201414
Record Dates: First submitted 2020-09-03; First posted 2020-09-11 (Actual); Results first posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Wound Heal
Keywords: Mohs surgery; Manuka honey; Secondary intention wound healing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- APIS Biomaterial on the Head (Experimental): Participants in this group will receive the experimental APIS Biomaterial on the Head. One layer of APIS® will be applied to the post-operative wound covered by petrolatum impregnated gauze, a non-stick Telfa pad, gauze, and Opsite tape. The biomaterial will be reapplied if it is completely absorbed at follow up and the wound depth below the epithelial level.
  Interventions: Device: Participants in this group will receive the experimental APIS Biomaterial on the Head.
- APIS Biomaterial on the Lower Extremities (Experimental): Participants in this group will receive the experimental APIS Biomaterial on the Lower Extremities. One layer of APIS® will be applied to the post-operative wound covered by petrolatum impregnated gauze, a non-stick Telfa pad, gauze, and Opsite tape. The biomaterial will be reapplied if it is completely absorbed at follow up and the wound depth below the epithelial level.
  Interventions: Device: Participants in this group will receive the experimental APIS Biomaterial on the Lower Extremities.
- Standard Secondary Intention Healing on the Head (Active Comparator): Participants in this group will receive standard secondary intention wound healing post-operative care on the Head. Post-operative wound will heal via conventional secondary intention. Application of petrolatum impregnated gauze, a non-stick Telfa pad, gauze, and Opsite tape.
  Interventions: Other: Standard Secondary Intention Healing on the Head
- Standard Secondary Intention Healing on the Lower Extremities (Active Comparator): Participants in this group will receive standard secondary intention wound healing post-operative care on the Lower Extremities. Post-operative wound will heal via conventional secondary intention. Application of petrolatum impregnated gauze, a non-stick Telfa pad, gauze, and Opsite tape.
  Interventions: Other: Standard Secondary Intention Healing on the Lower Extremities

INTERVENTIONS:
Device: Participants in this group will receive the experimental APIS Biomaterial on the Head. — One layer of APIS® will be applied to the post-operative wound on the head covered by petrolatum impregnated gauze, a non-stick Telfa pad, gauze, and Opsite tape.
  Arms: APIS Biomaterial on the Head
Device: Participants in this group will receive the experimental APIS Biomaterial on the Lower Extremities. — One layer of APIS® will be applied to the post-operative wound on the lower extremities covered by petrolatum impregnated gauze, a non-stick Telfa pad, gauze, and Opsite tape.
  Arms: APIS Biomaterial on the Lower Extremities
Other: Standard Secondary Intention Healing on the Head — Participants in this group will receive standard secondary intention wound healing post-operative care on the Head. Post-operative wound will heal via conventional secondary intention. Application of petrolatum impregnated gauze, a non-stick Telfa pad, gauze, and Opsite tape.
  Arms: Standard Secondary Intention Healing on the Head
Other: Standard Secondary Intention Healing on the Lower Extremities — Participants in this group will receive standard secondary intention wound healing post-operative care on the Lower Extremities. Post-operative wound will heal via conventional secondary intention. Application of petrolatum impregnated gauze, a non-stick Telfa pad, gauze, and Opsite tape.
  Arms: Standard Secondary Intention Healing on the Lower Extremities

SUMMARY:
The purpose of this study is to elucidate if a novel biomaterial containing gelatin, manuka honey, and hydroxyapatite enhances secondary intention healing when compared to conventional secondary intention healing for surgical defects after Mohs micrographic surgery on the head and distal lower extremities (below the knee). This novel biomaterial has already been FDA cleared for surgical wounds.

DETAILED DESCRIPTION:
Secondary intention healing (SIH) is often underutilized and has several advantages compared to primary surgical repair. Wound care is minimal, bleeding and infection are rare, and risks associated with primary closure (e.g. hematoma, suture granuloma, graft or flap failure) are non-existent. Importantly, SIH facilitates surveillance of tumor recurrence, whereas flaps and grafts may bury residual tumor. When used in appropriate anatomical locations, SIH leads to high patient satisfaction. However, SIH requires regular wound care that can be cumbersome to patients.

Prior studies utilizing biologic dressings have shown patients report better quality of life during the post-operative period related to less pain, decreased dressing changes, and faster healing times. Biologic dressings provide an alternative to surgical autografts and eliminate the risks associated with graft harvesting (e.g. pain, infection, and scarring). For many patients, the cosmetic outcome following healing is important. However, cosmetic outcome with SIH is variable and depends on many factors, namely location (e.g. concavities favorable), skin laxity, and underlying musculature. Exuberant granulation tissue, hypopigmented and telangiectatic scars are the most frequent adverse cosmetic outcomes with SIH.

The novel biomaterial APIS® (SweetBio, Inc. Memphis, TN) is an advanced synthesis of gelatin, manuka honey, and hydroxyapatite bioengineered to protect wounds, manage exudate, and maintain a moist environment. It is FDA cleared (FDA number K1827250) for wound management across 9 indications including surgical wounds. It has been used successfully in a small case series of 8 patients for post-operative Mohs surgical wounds on the head and distal lower extremities. Time to complete re-epithelialization was 6 weeks (42 days), suggesting a reduction in healing time compared to standard SIH times for the leg and head of 127 and 57 days, respectively. Use of this novel biomaterial to enhance SIH is hypothesized to reduce healing times when compared to standard SIH wound care. This provides a useful option to aid SIH in sites like the lower legs, where healing can be prolonged due to intrinsic factors (e.g., cardiovascular disease, peripheral vascular disease, diabetes) or extrinsic factors (e.g., increased risk of surgical site infection following dermatologic surgery at sites below the knee).

Randomized, comparative studies evaluating augmented SIH compared to conventional SIH in dermatologic surgery are limited. This study aims to evaluate whether use of a novel biomaterial enhances SIH, particularly in shortening time to complete re-epithelialization. Patients undergoing Mohs micrographic surgery amenable to SIH on the head and distal lower extremities will be randomized into one of four groups (standard SIH or biomaterial APIS® enhanced SIH on the head or distal lower extremities). Patients will have regularly scheduled follow-up with questionnaires at each visit. The investigators aim to evaluate whether use of this novel biomaterial decreases complete re-epithelialization times, reduces infection rates, and improves cosmetic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Post-operative wounds following Mohs surgery on the head or distal lower extremities
* Single Mohs post-operative defect
* Post-operative wounds greater than 1cm in width
* Depth of defect at least to subcutaneous tissue
* Patients have the ability to provide their own wound care
* Agreeable to regularly scheduled follow-up visits and transmission of photos via HIPAA compliant Vanderbilt University Medical Center Box
* Patients are able to provide informed consent

Exclusion Criteria:

* Under 18 years of age
* Unable to provide informed consent
* Unable to understand oral and written English
* Post-operative wounds not appropriate for secondary intention healing
* Sensitivity or allergy to APIS® biomaterial including collagen and its derivatives, porcine-derived materials or honey
* Immunosuppressed and organ transplant patients
* Post-operative wounds superficial to subcutaneous tissue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna S Clayton, MD, Study Director — Vanderbilt University Medical Center Dermatology
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zitelli JA. Wound healing by secondary intention. A cosmetic appraisal. J Am Acad Dermatol. 1983 Sep;9(3):407-15. doi: 10.1016/s0190-9622(83)70150-7. PMID 6630602
- [Background] Zitelli JA. Secondary intention healing: an alternative to surgical repair. Clin Dermatol. 1984 Jul-Sep;2(3):92-106. doi: 10.1016/0738-081x(84)90031-2. No abstract available. PMID 6400321
- [Background] Donaldson MR, Coldiron BM. Scars after second intention healing. Facial Plast Surg. 2012 Oct;28(5):497-503. doi: 10.1055/s-0032-1325643. Epub 2012 Oct 1. PMID 23027216
- [Background] Stebbins WG, Gusev J, Higgins HW 2nd, Nelson A, Govindarajulu U, Neel V. Evaluation of patient satisfaction with second intention healing versus primary surgical closure. J Am Acad Dermatol. 2015 Nov;73(5):865-7.e1. doi: 10.1016/j.jaad.2015.07.019. No abstract available. PMID 26475539
- [Background] Chern PL, Baum CL, Arpey CJ. Biologic dressings: current applications and limitations in dermatologic surgery. Dermatol Surg. 2009 Jun;35(6):891-906. doi: 10.1111/j.1524-4725.2009.01153.x. Epub 2009 Apr 6. PMID 19397669
- [Background] Eaglstein WH, Iriondo M, Laszlo K. A composite skin substitute (graftskin) for surgical wounds. A clinical experience. Dermatol Surg. 1995 Oct;21(10):839-43. doi: 10.1111/j.1524-4725.1995.tb00709.x. PMID 7551738
- [Background] Yang YW, Ochoa SA. Use of Porcine Xenografts in Dermatology Surgery: The Mayo Clinic Experience. Dermatol Surg. 2016 Aug;42(8):985-91. doi: 10.1097/DSS.0000000000000804. PMID 27340740
- [Background] Mott KJ, Clark DP, Stelljes LS. Regional variation in wound contraction of mohs surgery defects allowed to heal by second intention. Dermatol Surg. 2003 Jul;29(7):712-22. doi: 10.1046/j.1524-4725.2003.29180.x. PMID 12828694
- [Background] Deutsch BD, Becker FF. Secondary healing of Mohs defects of the forehead, temple, and lower eyelid. Arch Otolaryngol Head Neck Surg. 1997 May;123(5):529-34. doi: 10.1001/archotol.1997.01900050085011. PMID 9158402
- [Background] Chetter IC, Oswald AV, McGinnis E, Stubbs N, Arundel C, Buckley H, Bell K, Dumville JC, Cullum NA, Soares MO, Saramago P. Patients with surgical wounds healing by secondary intention: A prospective, cohort study. Int J Nurs Stud. 2019 Jan;89:62-71. doi: 10.1016/j.ijnurstu.2018.09.011. Epub 2018 Sep 18. PMID 30343210
- [Background] McMurray SL, Wallace MM, Stebbins WG, Clayton AS. Use of a Novel Biomaterial to Enhance Secondary Intention Healing. Dermatol Surg. 2021 Jun 1;47(6):843-844. doi: 10.1097/DSS.0000000000002725. No abstract available. PMID 32804895
- [Background] Dixon AJ, Dixon MP, Askew DA, Wilkinson D. Prospective study of wound infections in dermatologic surgery in the absence of prophylactic antibiotics. Dermatol Surg. 2006 Jun;32(6):819-26; discussion 826-7. doi: 10.1111/j.1524-4725.2006.32167.x. PMID 16792648
- [Derived] Arnaud K, Wallace MM, Wheless LE, Stebbins WG, Clayton AS. Novel Biomaterial Containing Gelatin, Manuka Honey, and Hydroxyapatite Enhanced Secondary Intention Healing Versus Standard Secondary Intention Healing in Mohs Surgical Defects on the Head and Distal Lower Extremities-A Randomized Controlled Trial: Pilot Study. Dermatol Surg. 2023 Dec 1;49(12):1160-1164. doi: 10.1097/DSS.0000000000003924. Epub 2023 Aug 30. PMID 37647156

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 10/8/2020-1/27/2022 at Vanderbilt University Medical Center within the Department of Dermatology Mohs Surgical Unit.
Pre-assignment Details: Thirty-seven participants were enrolled in total: 16 to the lower extremity group and 21 to the head group.
Groups:
- APIS Biomaterial on the Head (Intervention Group): Participants received the experimental APIS biomaterial on the head. One layer of APIS biomaterial will be applied to the post-operative wound covered by petrolatum impregnated gauze, a non-stick Telfa pad, gauze, and Opsite tape. The biomaterial will be reapplied if it is completely absorbed at follow up and the wound depth below the epithelial level.
- Standard Secondary Intention Healing on the Head (Control Group); Standard Secondary Intention Healing on the Lower Extremities (Control Group): Participants in this group received standard secondary intention wound healing post-operative care on the head. Post-operative wound will heal via conventional secondary intention. Application of petrolatum impregnated gauze, a non-stick Telfa pad, gauze, and Opsite tape.
- APIS Biomaterial on the Lower Extremities (Intervention Group): Participants received the experimental APIS biomaterial on the lower extremities. One layer of APIS biomaterial will be applied to the post-operative wound covered by petrolatum impregnated gauze, a non-stick Telfa pad, gauze, and Opsite tape. The biomaterial will be reapplied if it is completely absorbed at follow up and the wound depth below the epithelial level.
Period: Overall Study
Arm/Group | APIS Biomaterial on the Head (Intervention Group) | Standard Secondary Intention Healing on the Head (Control Group) | APIS Biomaterial on the Lower Extremities (Intervention Group) | Standard Secondary Intention Healing on the Lower Extremities (Control Group)
Started | 11 | 10 | 8 | 8
Completed | 10 | 9 | 8 | 8
Not Completed | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Sixteen patients with surgical defects on the lower extremities amenable and conducive for SIH were randomized to intervention or control by block randomization. Subjects were randomized in a 1:1 ratio. Twenty-one patients with surgical defects on the head were randomized in the same manner.
Groups:
- APIS Biomaterial on the Lower Extremities (Intervention Group): Participants received the experimental APIS biomaterial on the distal lower extremities. One layer of APIS biomaterial will be applied to the post-operative wound covered by petrolatum impregnated gauze, a non-stick Telfa pad, gauze, and Opsite tape. The biomaterial will be reapplied if it is completely absorbed at follow up and the wound depth below the epithelial level.
- Standard Secondary Intention Healing on the Lower Extremities (Control Group): Participants in this group received standard secondary intention wound healing post-operative care on the distal lower extremities. Post-operative wound will heal via conventional secondary intention. Application of petrolatum impregnated gauze, a non-stick Telfa pad, gauze, and Opsite tape.
- Total: Total of all reporting groups
Arm/Group | APIS Biomaterial on the Head (Intervention Group) | Standard Secondary Intention Healing on the Head (Control Group) | APIS Biomaterial on the Lower Extremities (Intervention Group) | Standard Secondary Intention Healing on the Lower Extremities (Control Group) | Total
Number analyzed (Participants) | 11 | 10 | 8 | 8 | 37
Age, Continuous [Mean (Full Range); unit: years] | 68.5 [35 to 85] | 74.6 [58 to 85] | 67.7 [59 to 92] | 71.2 [60 to 86] | 70.6 [35 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 6 | 5 | 14
  Male | 8 | 10 | 2 | 3 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 10 | 8 | 8 | 37

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Wound Re-epithelialization on the Head
Description: Complete wound re-epithelialization is defined by epidermal regrowth covering entire post-operative defect. Patients will be seen in office 14 days post-operative, then every 14 days thereafter until complete re-epithelialization is achieved. Patients will also submit photos via Vanderbilt HIPAA compliant Box at regular follow-up intervals (post-operative day 7 then every 14 days thereafter until complete re-epithelialization is achieved). Time elapsed from surgery date to complete re-epithelialization will be noted in days.
  Time will be measured in days. Increased days indicates slower wound healing.
Time Frame: 14 days post-operative until complete re-epithelialization, approximately 5 months
Population: Of the 21 randomized in the head group, 11 were randomized to the intervention group and 10 to the control group. One participant from the intervention group, and one participant from the control group were lost to follow up before complete re-epithelialization was achieved.
Measure: Mean (Standard Deviation); unit: days
Groups:
- APIS Biomaterial on Head (Intervention Group): Participants received the experimental APIS biomaterial on the head. One layer of APIS biomaterial will be applied to the post-operative wound covered by petrolatum impregnated gauze, a non-stick Telfa pad, gauze, and Opsite tape. The biomaterial will be reapplied if it is completely absorbed at follow up and the wound depth below the epithelial level.
Arm/Group | APIS Biomaterial on Head (Intervention Group) | Standard Secondary Intention Healing on the Head (Control Group)
Number analyzed (Participants) | 10 | 9
days | 41.6 (14.7) | 43 (12.3)

2. Primary Outcome: Time to Complete Wound Re-epithelialization on the Lower Extremities
Description: as for outcome 1
Time Frame: 14 days post-operative until complete re-epithelialization, approximately 5 months
Population: Analysis of re-epithelialization of wounds of the lower extremities with standard secondary intention healing versus APIS biomaterial.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | APIS Biomaterial on the Lower Extremities | Standard Secondary Intention Healing on the Lower Extremities
Number analyzed (Participants) | 8 | 8
days | 49.5 (19.1) | 52.7 (20.1)

3. Secondary Outcome: Patient Self Reported Pain Score
Description: Patients self-reported their surgical site/wound pain during each 2-week follow-up visit via a questionnaire. Scores were collected from participants until complete wound re-epithelialization, which was approximately 5 months for each participant.
  Pain scale will range from 1 (no pain) to 10 (worst pain imaginable). These pain scores were then averaged amongst the participants included in each arm.
Time Frame: Baseline to complete wound re-epithelialization, approximately 5 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Standard Secondary Intention Healing on the Lower Extremities (Control Group): Participants in this group received standard secondary intention wound healing post-operative care on the lower extremities. Post-operative wound will heal via conventional secondary intention. Application of petrolatum impregnated gauze, a non-stick Telfa pad, gauze, and Opsite tape.
Arm/Group | APIS Biomaterial on Head (Intervention Group) | Standard Secondary Intention Healing on the Head (Control Group) | APIS Biomaterial on the Lower Extremities (Intervention Group) | Standard Secondary Intention Healing on the Lower Extremities (Control Group)
Number analyzed (Participants) | 10 | 9 | 8 | 8
score on a scale | 1.25 (0.46) | 2.62 (1.41) | 1.14 (0.38) | 1.29 (0.49)

4. Secondary Outcome: Number of Participants With at Least One Post-Operative Wound Infection
Description: Post-operative wounds will be assessed for infection at regularly scheduled follow-ups. Any clinically suspected infection (e.g. erythema, purulence, malodor) will be reported.
Time Frame: Baseline to complete re-epithelialization, approximately 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | APIS Biomaterial on Head (Intervention Group) | Standard Secondary Intention Healing on the Head (Control Group) | APIS Biomaterial on the Lower Extremities (Intervention Group) | Standard Secondary Intention Healing on the Lower Extremities (Control Group)
Number analyzed (Participants) | 10 | 9 | 8 | 8
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With at Least One Report of Post-operative Bleeding
Description: Patients will report any bleeding (yes/no) via questionnaires at regularly scheduled follow-up appointments.
Time Frame: Baseline to complete re-epithelialization, approximately 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | APIS Biomaterial on Head (Intervention Group) | Standard Secondary Intention Healing on the Head (Control Group) | APIS Biomaterial on the Lower Extremities (Intervention Group) | Standard Secondary Intention Healing on the Lower Extremities (Control Group)
Number analyzed (Participants) | 10 | 9 | 8 | 8
Participants | 1 | 2 | 0 | 0

6. Secondary Outcome: Skin Thickness
Description: Participants were given a questionnaire at the final visit when complete wound re-epithelialization had been achieved (which was approximately 5 months for each participant) and asked, "Is the thickness of the scar different from your normal skin at present?" Participants reported on a scale of 1 (no, as normal skin) to 10 (yes, very different). These skin thickness scores were then averaged amongst the participants included in each arm.
Time Frame: Baseline to complete wound re-epithelialization, approximately 5 months
Population: Two patients in the intervention group for the head, 2 patients in control group for the head, 1 patient in intervention group for lower extremities and 1 patient in control group for lower extremities failed to complete a final questionnaire on scar assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | APIS Biomaterial on Head (Intervention Group) | Standard Secondary Intention Healing on the Head (Control Group) | APIS Biomaterial on the Lower Extremities (Intervention Group) | Standard Secondary Intention Healing on the Lower Extremities (Control Group)
Number analyzed (Participants) | 8 | 7 | 7 | 7
score on a scale | 2.38 (0.74) | 6.5 (1.77) | 4.43 (1.81) | 3.29 (1.60)

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for the study.
Arm/Group | APIS Biomaterial on the Head | APIS Biomaterial on the Lower Extremities | Standard Secondary Intention Healing on the Head | Standard Secondary Intention Healing on the Lower Extremities
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
It was difficult to enroll patients during the COVID-19 pandemic as regular follow up visits were required.

Of the 21 patients enrolled in the head group, two were lost to follow up. The low infection rate could possibly be attributed to patients with defects on the distal lower extremities receiving prophylactic antibiotics. Photos taken at follow-up visits were not taken in standardized format, so the difference in wound healing may not be as evident photographically as it was clinically.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT04545476/Prot_SAP_000.pdf